CLINICAL TRIAL: NCT02955394
Title: Randomized Phase II Trial of Preoperative Fulvestrant With or Without Enzalutamide in ER+/Her2- Breast Cancer
Brief Title: Preoperative Fulvestrant With or Without Enzalutamide in ER+/Her2- Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1042.cc
Record Dates: First submitted 2016-11-01; First posted 2016-11-04 (Estimated); Results first posted 2023-06-15 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: ER+/Her2 - breast cancer; Preoperative Fulvestrant; Enzalutamide
MeSH Terms: conditions — Breast Neoplasms | interventions — enzalutamide; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fulvestrant Without Enzalutamide (Placebo Comparator): 500 mg of Fulvestrant will be given IM on days 1, 15, 28, then every 4 weeks as per standard of care (SOC)
  Interventions: Drug: Fulvestrant
- Fulvestrant With Enzalutamide (Experimental): 500 mg of Fulvestrant will be given IM on days 1, 15, 28, then every 4 weeks as per standard of care (SOC), plus160mg of Enzalutamide will be given daily.
  Interventions: Drug: Enzalutamide; Drug: Fulvestrant

INTERVENTIONS:
Drug: Enzalutamide — 160mg of Enzalutamide will be given daily in conjunction with Fulvestrant.
  Other Names: MDV3100
  Arms: Fulvestrant With Enzalutamide
Drug: Fulvestrant — 500mg Fulvestrant will be given IM on days 1, 15, 28, then every 4 weeks as per standard of care (SOC)
  Other Names: FASLODEX

SUMMARY:
This is a randomized two arm phase II study to further evaluate the efficacy of fulvestrant plus enza compared to single agent fulvestrant in postmenopausal women with locally advanced AR+/ER+/Her2- BC who will have local surgery after ~4 months on treatment.

DETAILED DESCRIPTION:
This is a randomized two arm phase II study to further evaluate the efficacy of fulvestrant plus enza compared to single agent fulvestrant in postmenopausal women with locally advanced AR+/ER+/Her2- BC who will have local surgery after ~4 months on treatment. After consent, all patients will get a tissue biopsy, and than half the patients will get fulvestrant alone (standard dosing) and the other half of the patients will get fulvestrant plus enzalutamide. At ~4 weeks, a biopsy will be done and therapy will be continued. Hormone therapy will continue for ~4 months at which point the patients will undergo surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* ER+ Her2- breast cancer
* Stage at least T2 or greater
* Planned to get local surgery
* Postmenopausal, or if pre- or peri- menopausal, then will need to have concurrent ovarian suppression.
* At least 18 years of age
* Not on anticoagulants
* PS 0-2
* Able to swallow study drug and comply with study requirements
* ANC >1000/uL, platelets >75,000/uL at screening visit
* Total bilirubin < 1.5 times upper limit of normal (ULN) at the screening visit unless an alternate nonmalignant etiology exists (eg, Gilbert's disease)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 3 times ULN or < 5 times ULN if patient has documented liver metastases
* Creatinine < 1.5 times ULN
* INR < 1.5 times ULN, or if on warfarin, can safely transition off for biopsy
* Willing to donate blood for research at 4 time points
* Willing to undergo core biopsies for research at study entry and at ~4 weeks.
* Willing to donate tissue to research from the surgical specimen
* Written informed consent obtained prior to biopsies and blood samples

Exclusion Criteria:

* Current or previously treated brain or leptomeningeal metastases
* History of seizures
* Prior treatment with an anti-androgen (abiraterone, ARN-509, bicalutamide, enzalutamide, ODM-201, TAK-448, TAK-683, TAK-700, VT-464).
* Systemic estrogens or androgens within 14 days before initiating therapy. Vaginal estrogens are allowed if necessary for patient comfort.

Ages: 18 Years to 101 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2027-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony D Elias, MD, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - University of Colorado, Aurora, Colorado
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - West Cancer Center, Germantown, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Collins LC, Cole KS, Marotti JD, Hu R, Schnitt SJ, Tamimi RM. Androgen receptor expression in breast cancer in relation to molecular phenotype: results from the Nurses' Health Study. Mod Pathol. 2011 Jul;24(7):924-31. doi: 10.1038/modpathol.2011.54. Epub 2011 May 6. PMID 21552212
- [Background] Elebro K, Borgquist S, Simonsson M, Markkula A, Jirstrom K, Ingvar C, Rose C, Jernstrom H. Combined Androgen and Estrogen Receptor Status in Breast Cancer: Treatment Prediction and Prognosis in a Population-Based Prospective Cohort. Clin Cancer Res. 2015 Aug 15;21(16):3640-50. doi: 10.1158/1078-0432.CCR-14-2564. Epub 2015 Apr 22. PMID 25904752
- [Background] Hu R, Dawood S, Holmes MD, Collins LC, Schnitt SJ, Cole K, Marotti JD, Hankinson SE, Colditz GA, Tamimi RM. Androgen receptor expression and breast cancer survival in postmenopausal women. Clin Cancer Res. 2011 Apr 1;17(7):1867-74. doi: 10.1158/1078-0432.CCR-10-2021. Epub 2011 Feb 15. PMID 21325075
- [Background] Cochrane DR, Bernales S, Jacobsen BM, Cittelly DM, Howe EN, D'Amato NC, Spoelstra NS, Edgerton SM, Jean A, Guerrero J, Gomez F, Medicherla S, Alfaro IE, McCullagh E, Jedlicka P, Torkko KC, Thor AD, Elias AD, Protter AA, Richer JK. Role of the androgen receptor in breast cancer and preclinical analysis of enzalutamide. Breast Cancer Res. 2014 Jan 22;16(1):R7. doi: 10.1186/bcr3599. PMID 24451109
- [Background] D'Amato NC, Gordon MA, Babbs B, Spoelstra NS, Carson Butterfield KT, Torkko KC, Phan VT, Barton VN, Rogers TJ, Sartorius CA, Elias A, Gertz J, Jacobsen BM, Richer JK. Cooperative Dynamics of AR and ER Activity in Breast Cancer. Mol Cancer Res. 2016 Nov;14(11):1054-1067. doi: 10.1158/1541-7786.MCR-16-0167. Epub 2016 Aug 26. PMID 27565181
- [Background] Takagi K, Miki Y, Nagasaki S, Hirakawa H, Onodera Y, Akahira J, Ishida T, Watanabe M, Kimijima I, Hayashi S, Sasano H, Suzuki T. Increased intratumoral androgens in human breast carcinoma following aromatase inhibitor exemestane treatment. Endocr Relat Cancer. 2010 Apr 21;17(2):415-30. doi: 10.1677/ERC-09-0257. Print 2010 Jun. PMID 20228125
- [Background] Elias A, Richer JK, LoRusso P, Peterson AC, Steinberg J, Mordenti J, Lopez C, Hudis C, Traina T. MDV3100-08: A phase 1 open-label, dose-escalation study evaluating the safety, tolerability, and pharmacokinetics of MDV3100 in women with incurable breast cancer. ASCO 2012, TPS668
- [Background] Scher HI, Fizazi K, Saad F, Taplin ME, Sternberg CN, Miller K, de Wit R, Mulders P, Chi KN, Shore ND, Armstrong AJ, Flaig TW, Flechon A, Mainwaring P, Fleming M, Hainsworth JD, Hirmand M, Selby B, Seely L, de Bono JS; AFFIRM Investigators. Increased survival with enzalutamide in prostate cancer after chemotherapy. N Engl J Med. 2012 Sep 27;367(13):1187-97. doi: 10.1056/NEJMoa1207506. Epub 2012 Aug 15. PMID 22894553
- [Background] Yeo B, Dowsett M. Neoadjuvant endocrine therapy: Patient selection, treatment duration and surrogate endpoints. Breast. 2015 Nov;24 Suppl 2:S78-83. doi: 10.1016/j.breast.2015.07.019. Epub 2015 Aug 6. PMID 26255746
- [Background] Charehbili A, Fontein DB, Kroep JR, Liefers GJ, Mieog JS, Nortier JW, van de Velde CJ. Neoadjuvant hormonal therapy for endocrine sensitive breast cancer: a systematic review. Cancer Treat Rev. 2014 Feb;40(1):86-92. doi: 10.1016/j.ctrv.2013.06.001. Epub 2013 Jul 23. PMID 23891267
- [Background] Semiglazov VF, Semiglazov VV, Dashyan GA, Ziltsova EK, Ivanov VG, Bozhok AA, Melnikova OA, Paltuev RM, Kletzel A, Berstein LM. Phase 2 randomized trial of primary endocrine therapy versus chemotherapy in postmenopausal patients with estrogen receptor-positive breast cancer. Cancer. 2007 Jul 15;110(2):244-54. doi: 10.1002/cncr.22789. PMID 17538978
- [Background] von Minckwitz G, Untch M, Nuesch E, Loibl S, Kaufmann M, Kummel S, Fasching PA, Eiermann W, Blohmer JU, Costa SD, Mehta K, Hilfrich J, Jackisch C, Gerber B, du Bois A, Huober J, Hanusch C, Konecny G, Fett W, Stickeler E, Harbeck N, Muller V, Juni P. Impact of treatment characteristics on response of different breast cancer phenotypes: pooled analysis of the German neo-adjuvant chemotherapy trials. Breast Cancer Res Treat. 2011 Jan;125(1):145-56. doi: 10.1007/s10549-010-1228-x. Epub 2010 Nov 3. PMID 21042932
- [Background] Kaufmann M, Hortobagyi GN, Goldhirsch A, Scholl S, Makris A, Valagussa P, Blohmer JU, Eiermann W, Jackesz R, Jonat W, Lebeau A, Loibl S, Miller W, Seeber S, Semiglazov V, Smith R, Souchon R, Stearns V, Untch M, von Minckwitz G. Recommendations from an international expert panel on the use of neoadjuvant (primary) systemic treatment of operable breast cancer: an update. J Clin Oncol. 2006 Apr 20;24(12):1940-9. doi: 10.1200/JCO.2005.02.6187. PMID 16622270
- [Background] Dowsett M, Smith IE, Ebbs SR, Dixon JM, Skene A, Griffith C, Boeddinghaus I, Salter J, Detre S, Hills M, Ashley S, Francis S, Walsh G; IMPACT Trialists. Short-term changes in Ki-67 during neoadjuvant treatment of primary breast cancer with anastrozole or tamoxifen alone or combined correlate with recurrence-free survival. Clin Cancer Res. 2005 Jan 15;11(2 Pt 2):951s-8s. PMID 15701892
- [Background] Ellis MJ, Ma C. Letrozole in the neoadjuvant setting: the P024 trial. Breast Cancer Res Treat. 2007;105 Suppl 1(Suppl 1):33-43. doi: 10.1007/s10549-007-9701-x. Epub 2007 Oct 3. PMID 17912634
- [Background] Ellis MJ, Llombart-Cussac A, Feltl D, Dewar JA, Jasiowka M, Hewson N, Rukazenkov Y, Robertson JF. Fulvestrant 500 mg Versus Anastrozole 1 mg for the First-Line Treatment of Advanced Breast Cancer: Overall Survival Analysis From the Phase II FIRST Study. J Clin Oncol. 2015 Nov 10;33(32):3781-7. doi: 10.1200/JCO.2015.61.5831. Epub 2015 Sep 14. PMID 26371134
- [Background] Robertson JF, Lindemann JP, Llombart-Cussac A, Rolski J, Feltl D, Dewar J, Emerson L, Dean A, Ellis MJ. Fulvestrant 500 mg versus anastrozole 1 mg for the first-line treatment of advanced breast cancer: follow-up analysis from the randomized 'FIRST' study. Breast Cancer Res Treat. 2012 Nov;136(2):503-11. doi: 10.1007/s10549-012-2192-4. Epub 2012 Oct 13. PMID 23065000
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Derived] Elias AD, Staley AW, Fornier M, Vidal GA, Alami V, Sams S, Spoelstra NS, Goodspeed A, Kabos P, Diamond JR, Shagisultanova E, Gallagher RI, Wulfkuhle JD, Petricoin EF, Zolman KL, McSpadden T, Jordan KR, Slansky JE, Borges VF, Gao D, Richer JK. Clinical and immune responses to neoadjuvant fulvestrant with or without enzalutamide in ER+/Her2- breast cancer. NPJ Breast Cancer. 2024 Oct 6;10(1):88. doi: 10.1038/s41523-024-00697-5. PMID 39368973

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fulvestrant Without Enzalutamide | Fulvestrant With Enzalutamide
Started | 27 | 34
Completed | 25 | 32
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fulvestrant Without Enzalutamide | Fulvestrant With Enzalutamide | Total
Number analyzed (Participants) | 27 | 34 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 9 | 15 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (13.08) | 61.47 (10.10) | 60.49 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 34 | 61
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 27 | 32 | 59
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 10 | 12
  White | 22 | 24 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 27 | 34 | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a PEPI Score Equal to Zero at Post Treatment
Description: The preoperative endocrine prognostic index (PEPI) is a validated measure of pathologic response to endocrine therapy. It is a model that combines estrogen receptor (ER) level, pathologic tumor site, nodal status, and Ki67 score at the time of surgery to predict subsequent risk of cancer recurrence.
  PEPI scoring is typically discretized into three risk groups: 0 (low risk of recurrence and best outcome), 1-3 (intermediate risk), and >= 4 (high risk). This study was concerned only with the distinction between zero and non-zero PEPI scores. Zero is the minimum score, and there is no maximum score. Lower scores are better.
Time Frame: 16 Weeks
Population: 59 patients were evaluable. One patient was unable to participate in treatment after baseline and the other came off study for treatment change.
Measure: Count of Participants; unit: Participants
Arm/Group | Fulvestrant Without Enzalutamide | Fulvestrant With Enzalutamide
Number analyzed (Participants) | 26 | 33
Participants | 2 | 8

2. Secondary Outcome: Disease-free Survival
Description: Disease-free survival is defined as the time in months from the start of fulvestrant until documented disease progression or death. Complete and partial response for the single drug arm and combination of enzalutamide/fulvestrant arm separately.
Time Frame: 15 months
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Fulvestrant Without Enzalutamide | Fulvestrant With Enzalutamide
Number analyzed (Participants) | 26 | 33
months | 3.6 [2.5 to 5.8] | 3.7 [0.9 to 15.2]

3. Secondary Outcome: Correlation Between PEPI Score and Disease-free Survival, Clinical Benefit Rate, and Overall Response Rate
Description: To assess the association between PEPI score and the clinical, outcomes such as DFS, ORR, clinical benefit for all subjects.
Time Frame: 4 years
Reporting Status: Not Posted

4. Secondary Outcome: Androgen Receptor (AR) Expression
Description: The strength of AR signaling was measured by the percentage of downstream AR-regulated genes that were expressed.
Time Frame: 16 Weeks
Population: The number of evaluable patients for this outcome measure is 49 because these were the patients who had available lab data for AR%.
Measure: Median (Full Range); unit: percentage of genes expressed
Arm/Group | Fulvestrant Without Enzalutamide | Fulvestrant With Enzalutamide
Number analyzed (Participants) | 22 | 27
percentage of genes expressed | 85 [10 to 100] | 80 [10 to 100]

ADVERSE EVENTS:
Time Frame: 51.78 months
Arm/Group | Fulvestrant Without Enzalutamide | Fulvestrant With Enzalutamide
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/34
Serious Adverse Events (participants affected / at risk) | 1/27 | 3/34
Other Adverse Events (participants affected / at risk) | 26/27 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant Without Enzalutamide (N=27) | Fulvestrant With Enzalutamide (N=34)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant Without Enzalutamide (N=27) | Fulvestrant With Enzalutamide (N=34)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (2) | 2 (2)
Alanine Aminotransferase Increased (Hepatobiliary disorders) | 1 (2) | 1 (1)
Alkaline Phosphatase Increase (Hepatobiliary disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 4 (4)
Arthralgia (Immune system disorders) | 4 (4) | 5 (5)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 1 (1) | 3 (3)
Cognitive Disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 4 (4)
Creatinine increased (Renal and urinary disorders) | 1 (2) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 9 (11)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 8 (10) | 17 (24)
Abdominal Cramping (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 3 (3) | 14 (21)
Hot flashes (Vascular disorders) | 12 (12) | 13 (19)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Papular Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 13 (14)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2)
Weight Gain (Investigations) | 1 (1) | 1 (1)
decreased activity (General disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 7 (9) | 16 (18)
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pain (General disorders) | 6 (8) | 13 (17)
Paresthesia (Nervous system disorders) | 2 (2) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Maculo-papular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Seroma (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
tremor (Nervous system disorders) | 1 (1) | 2 (2)
Skin disorders (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (7)
Urinary issues (Renal and urinary disorders) | 1 (1) | 1 (1)
vaginal dryness (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 4 (10)
alanine transaminase increase (Investigations) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blurred Vision (Eye disorders) | 0 (0) | 2 (3)
agitation (Psychiatric disorders) | 0 (0) | 2 (2)
Anorgasmia (Psychiatric disorders) | 0 (0) | 1 (1)
Edema (General disorders) | 0 (0) | 2 (2)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
Concentration Impairment (Nervous system disorders) | 0 (0) | 3 (4)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 5 (5)
Dizziness (Nervous system disorders) | 0 (0) | 6 (8)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (2)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (6)
Euphoria (Psychiatric disorders) | 0 (0) | 1 (1)
Eye disorders (Eye disorders) | 0 (0) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0)
Hypertension (Surgical and medical procedures) | 0 (0) | 2 (2)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Loss of Taste (Investigations) | 0 (0) | 1 (1)
Muscle pain (Investigations) | 0 (0) | 1 (1)
Restless Leg Syndrome (Investigations) | 0 (0) | 1 (1)
Cold intolerance (General disorders) | 0 (0) | 1 (1)
Neck tightness (General disorders) | 0 (0) | 1 (1)
restless hands (General disorders) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
Increase Urine Output (Renal and urinary disorders) | 0 (0) | 2 (2)
Decreased ROM (General disorders) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Decreased libido (Psychiatric disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Weight Loss (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Pre-Diabeties (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Appetite Change (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Involuntary movement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 0 (0) | 3 (3)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nervous System Disorders (Nervous system disorders) | 0 (0) | 6 (8)
Oral Hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Peripheral Sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Personality Change (Psychiatric disorders) | 0 (0) | 1 (1)
postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Vaginal Bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Respiratory issues (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (7)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Toothache (General disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Vaginal Discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal Infection (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT02955394/Prot_SAP_ICF_001.pdf